CLINICAL TRIAL: NCT04536896
Title: Efficacy of a Smartphone App for a Breastmilk Feeding Course Among Sixth Year Medical Students
Brief Title: Smartphone Application for Breastfeeding Education in Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Erika Ochoa-Correa, Medical Doctor, Universidad Autonoma de Nuevo Leon
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PE18-00005
Record Dates: First submitted 2020-08-22; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Medical Education
Keywords: breastfeeding education; medical education

STUDY DESIGN:
Intervention Model Description: Non-randomized quasi-experimental trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional face-to-face teaching method (Active Comparator): In this arm, participants underwent a 6-hour traditional face-to-face lecture on breastfeeding education in a classroom at a university. Course was divided into 4 1.5-hour sessions during a time span of two weeks.
  Interventions: Other: Traditional face-to-face breastfeeding lecture
- Breastfeeding smartphone app (Experimental): In this group, participants downloaded a smartphone application which contained an online breastfeeding education course. Participants freely navigated through the smartphone app during a time span of two weeks.
  Interventions: Other: Smartphone breastfeeding application

INTERVENTIONS:
Other: Smartphone breastfeeding application — This intervention consists of a smartphone application which contains relevant information and topics regarding proper breastfeeding knowledge for medical students.
  Arms: Breastfeeding smartphone app
Other: Traditional face-to-face breastfeeding lecture — This intervention consists of the impartition of a face-to-face breastfeeding course
  Arms: Traditional face-to-face teaching method

SUMMARY:
The purpose of this study was to compare the efficacy of two educational interventions to enhance breastfeeding knowledge among senior medical students. One intervention consisted of a traditional face-to-face teaching lecture and the other consisted of the use of a smartphone application containing information about breastfeeding.

DETAILED DESCRIPTION:
A quasi-experimental study was performed. Students were allocated to two groups; the first group underwent a 6-hour face-to-face breastfeeding course which was divided in four 1.5-hour sessions during a time span of two weeks. The second intervention consisted of downloading a digital smartphone application designed by the research team to teach proper breastfeeding concepts which participants freely navigated during the same time span of two weeks. Before and after each intervention, students answered a general breastfeeding knowledge test consisting of twenty multiple choice answers with a score range of 0 to 20. Statistical comparisons between pre- and post-test scores were performed in each group and mean change in scores was compared between them to establish which method was the most efficient. Moreover, amount of time spent on the application was descriptively measured.

ELIGIBILITY:
Inclusion Criteria:

* Senior adult medical students of any gender who at the time were enrolled on the Pediatrics biannual course during the July 2018 th -July 2019 th academic period.
* Provide verbal informed consent
* At least 18 years old

Exclusion Criteria:

* Students who did not possess an electronic device (smartphone or tablet) or decided not to participate in the study.
* Rate of non-attendance to the general pediatric course greater than 50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of each breastfeeding course evaluated by a quantitative general knowledge questionnaire | 14 days
  In order to measure this outcome, all participants answered a test consisting of a quantitative questionnaire of general breastfeeding knowledge before and after the intervention. This general knowledge test consisted of twenty questions with multiple choice answers ranging between two to five possible answers according to the nature of the question. It was designed by study researchers which included specialists in Pediatrics and breastfeeding and it was based solely on the course content. Minimum and maximum scores were 0 and 20, where a higher score indicated a better grade on the test. Central tendency and dispersion measures were obtained for pre- and post-test scores and a further statistical comparison between this parameters indicated whether there was a statistically significant difference. If the post-test score was statistically superior to the pre-test score, it was concluded that the intervention was efficient to improve breastfeeding knowledge.

SECONDARY OUTCOMES:
Comparison of the efficacy of each breastfeeding course by comparison of mean differences | 14 days
  In order to measure this outcome, a mean difference between the post-test and pre-test scores was obtained for each group. Furthermore, these mean differences were compared to establish if the mean improvement in test scores was different between both interventions. If the mean change of one intervention was statistically superior to the other, it was assumed that the former intervention was more efficient to promote breastfeeding knowledge. On the contrary, if no statistical differences between the effects of both interventions on test scores were observed, it was assumed that no intervention was superior to the other.
Amount of time in minutes spent on the smartphone application | 14 days
  Study researchers had access to the amount of time in minutes that each student dedicated to studying on the smartphone application. Descriptive statistics with central and dispersion tendencies were obtained to evaluate this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Ochoa-Correa, MD, Principal Investigator — UNIVERSIDAD AUTONOMA DE NUEVO LEON, School of Medicine, Department of Pediatrics
Locations (1):
- Facultad de Medicina, Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No
At request of other researchers, sharing of IPD will be assessed by the research team assuring confidentiality of participants information.

REFERENCES:
- [Background] Brudenell I, Carpenter CS. Adult learning styles and attitudes toward computer assisted instruction. J Nurs Educ. 1990 Feb;29(2):79-83. doi: 10.3928/0148-4834-19900201-08. PMID 2154567
- [Background] Lynch TG, Steele DJ, Johnson Palensky JE, Lacy NL, Duffy SW. Learning preferences, computer attitudes, and test performance with computer-aided instruction. Am J Surg. 2001 Apr;181(4):368-71. doi: 10.1016/s0002-9610(01)00575-x. PMID 11438276
- [Background] Davidson LK. A 3-year experience implementing blended TBL: active instructional methods can shift student attitudes to learning. Med Teach. 2011;33(9):750-3. doi: 10.3109/0142159X.2011.558948. Epub 2011 May 19. PMID 21592018
- [Background] Krupat E, Richards JB, Sullivan AM, Fleenor TJ Jr, Schwartzstein RM. Assessing the Effectiveness of Case-Based Collaborative Learning via Randomized Controlled Trial. Acad Med. 2016 May;91(5):723-9. doi: 10.1097/ACM.0000000000001004. PMID 26606719
- [Background] Anjum Q, Ashfaq T, Siddiqui H. Knowledge regarding breastfeeding practices among medical students of Ziauddin University Karachi. J Pak Med Assoc. 2007 Oct;57(10):480-3. PMID 17990420
- [Background] Freed GL, Clark SJ, Sorenson J, Lohr JA, Cefalo R, Curtis P. National assessment of physicians' breast-feeding knowledge, attitudes, training, and experience. JAMA. 1995 Feb 8;273(6):472-6. doi: 10.1001/jama.1995.03520300046035. PMID 7837365
- [Background] Silvestre PK, Carvalhaes MA, Venancio SI, Tonete VL, Parada CM. Breastfeeding knowledge and practice of health professionals in public health care services. Rev Lat Am Enfermagem. 2009 Nov-Dec;17(6):953-60. doi: 10.1590/s0104-11692009000600005. PMID 20126936
- [Background] de Almeida JM, Luz Sde A, Ued Fda V. [Support of breastfeeding by health professionals: integrative review of the literature]. Rev Paul Pediatr. 2015 Jul-Sep;33(3):356-63. doi: 10.1016/j.rpped.2014.10.002. Epub 2015 Jun 10. PMID 26141902
- [Background] Arthur CR, Saenz RB, Replogle WH. Personal breast-feeding behaviors of female physicians in Mississippi. South Med J. 2003 Feb;96(2):130-5. doi: 10.1097/01.SMJ.0000051268.43410.45. PMID 12630635
- [Background] Hall Moran V, Edwards J, Dykes F, Downe S. A systematic review of the nature of support for breast-feeding adolescent mothers. Midwifery. 2007 Jun;23(2):157-71. doi: 10.1016/j.midw.2006.06.005. Epub 2006 Oct 18. PMID 17052824
- [Background] Dykes F. The education of health practitioners supporting breastfeeding women: time for critical reflection. Matern Child Nutr. 2006 Oct;2(4):204-16. doi: 10.1111/j.1740-8709.2006.00071.x. PMID 16999766
- [Background] Caminha Mde F, Serva VB, dos Anjos MM, Brito RB, Lins MM, Batista Filho M. [Exclusive breastfeeding among professionals in a Family Healthcare Program]. Cien Saude Colet. 2011 Apr;16(4):2245-50. doi: 10.1590/s1413-81232011000400023. Portuguese. PMID 21584465
- [Background] Hoddinott P, Pill R, Chalmers M. Health professionals, implementation and outcomes: reflections on a complex intervention to improve breastfeeding rates in primary care. Fam Pract. 2007 Feb;24(1):84-91. doi: 10.1093/fampra/cml061. Epub 2006 Dec 7. PMID 17158185
- [Background] Yang SF, Salamonson Y, Burns E, Schmied V. Breastfeeding knowledge and attitudes of health professional students: a systematic review. Int Breastfeed J. 2018 Feb 20;13:8. doi: 10.1186/s13006-018-0153-1. eCollection 2018. PMID 29483935
- [Background] Gary AJ, Birmingham EE, Jones LB. Improving breastfeeding medicine in undergraduate medical education: A student survey and extensive curriculum review with suggestions for improvement. Educ Health (Abingdon). 2017 May-Aug;30(2):163-168. doi: 10.4103/efh.EfH_180_15. PMID 28928347